CLINICAL TRIAL: NCT00511563
Title: A Double-blind, Randomised, Placebo-controlled, Three-period Crossover Study to Investigate the Pharmacodynamic Effect of Two CRF-1 Antagonists GSK561679 and GW876008 on Meal Induced Cortisol Responses in Patients With IBS.
Brief Title: A Study In Patients With Irritable Bowel Syndrome To Measure Hormone Response After Dosing With GW876008 And Gsk561679
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Cancelled before active due to the results of emerging scientific data
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRI109244
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Cortisol,; stress,; response,; Irritable Bowel Syndrome,; cytokine.
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — GW 876008; NBI 77860

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- GW876008 and GSK561679 (Experimental): GW876008 and GSK561679
  Interventions: Drug: GW876008 and GSK561679

INTERVENTIONS:
Drug: GW876008 and GSK561679 — GW876008 and GSK561679

SUMMARY:
To better understand the way that GW876008 and GSK561679 work on hormone responses in patients with Irritable Bowel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Has IBS as defined by the Rome II criteria.
* Clinical laboratory tests at screening showing no clinically significant abnormalities in the opinion of the Principal Investigator.
* Non-tobacco user (abstinence from tobacco use for at least 1 month before the start of the study).

Exclusion Criteria:

* As a result of any of the medical interview, physical examination, evaluation of mental state and psychiatric history or screening investigations the physician responsible considers the subject unfit for the study.
* Subject has any of the following exclusionary psychiatric conditions (Note: current diagnoses are to be based on the M.I.N.I administered at screening).
* 1. A current DSM-IV Axis I disorder such as Dysthymia, Phobia, Major Depression, Obsessive Compulsive Disorder, Body Dysmorphic disorder, or Panic Disorder as a primary diagnosis currently or within 6 months prior to the screening visit.
* 2. A current DSM-IV-TR diagnosis of Antisocial or Borderline Personality Disorder, Dementia, or another current DSM-IV-TR Axis II diagnosis that would suggest non-responsiveness to pharmacotherapy or non-compliance with the protocol; or
* 3. A current (within six months prior to Screening Visit) diagnosis of anorexia nervosa or bulimia; or
* 4. A history of Schizophrenia, Schizoaffective Disorder, or a Bipolar Disorder; or
* 5. Is currently being treated by medication for any of the above psychiatric disorders. Psychiatric medications would include, but not limited to, antidepressants (e.g. SSRIs, SNRIs, TCAs) anxiolytics, antipsychotics
* Subjects who, in the investigator's judgement, pose a current, serious or suicidal or homicidal risk or have made a suicide attempt within the past 6 months or have ever been homicidal.
* subjects who have taken any medication for the treatment of IBS within 1 month prior to screening except for anti-diarrhoeal medications or laxatives for control of bowel habit which is allowed if at a stable dose for 2 weeks prior to randomisation.
* Subjects who are taking NSAIDs including aspirin on a regular basis or within 48 hours of a study day.
* Subjects with a history of PUD <10 years ago.
* The subject has a history of, or active eating disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Serum cortisol / ACTH and DHEA levels | taken at 20 minute intervals over the study period.

SECONDARY OUTCOMES:
Serum cytokine levels | taken at 20 minute intervals over the study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline